CLINICAL TRIAL: NCT01923051
Title: Czech Multicentre Research Database of Chronic Obstructive Pulmonary Disease (COPD): Registry of the Czech Pneumological Society (CPPS) at the Czech Medical Association (CzMA)
Brief Title: Czech Multicentre Research Database of Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zuzana Zbožínková, M.Sc. (Other)
Responsible Party: Sponsor-Investigator, Zuzana Zbožínková, M.Sc., Zuzana Zbozinkova PharmDr, Masaryk University
Organization: Masaryk University (Other)
Other Study IDs: 1301100001; 1301100001 (Other: State Institute for Drug Control, Czech Republic)
Record Dates: First submitted 2013-08-07; First posted 2013-08-14 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Airway Disease
Keywords: chronic obstructive pulmonary disease; COPD; national database; observational
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In the following centres, we will be collecting samples with DNA (blood samples): University Hospital Olomouc, University Hospital Hradec Kralove, University Hospital Motol, University Hospital Brno.
Oversight: Data Monitoring Committee: No

SUMMARY:
The chronic obstructive pulmonary disease (COPD) is the occurrence of chronic bronchitis or emphysema, a pair of commonly co-existing diseases of the lungs in which the airways narrow over time. This limits airflow to and from the lungs, causing shortness of breath (dyspnoea). In clinical practice, COPD is defined by its characteristic airflow limitation on lung function tests. In contrast to asthma, this limitation is poorly reversible and usually gets increasingly worse over time.

The COPD registry is a non-interventional multicentre observational prospective database focusing on the collection and analysis of data on real mortality and morbidity in COPD population of the Czech Republic population of COPD patients. Monitoring is done at the occasion of regular check-ups, followed by retrospective search of data in the documentation, and a record into the registry.

The aim of Czech National Research Database of Chronic Obstructive Pulmonary Disease is to establish the clinical course of severe forms of COPD, establish the cause for deterioration of clinical status of our patients and describe the progression of COPD to death.

The registry fulfils general objectives of health registries such as monitoring of causes, development, treatment and consequences of a severe disorder, including economic and social impacts. Statistical and scientific analyses of the registry data are focused, in particular, on the assessment of health determiners of the selected patient cohort with the aim to improve health status of the patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a treatable and preventable clinically heterogeneous syndrome with dominant respiratory symptoms and various systemic consequences. The incidence of COPD is increasing worldwide. In general, COPD is caused by a prolonged inflammatory reaction of a genetically predisposed individual exposed to long-term inhalation of air pollution, harmful particles and gases. This disease has a negative progression in time even after end of exposure. The pulmonary component is associated with expiratory airflow limitation, which is not fully reversible. The airflow limitation in COPD develops gradually as a result of chronic, primarily non-infectious inflammation of the airways and lung parenchyma. Systemic consequences are often found in cardiovascular, musculoskeletal and other systems. COPD can be considered a proven pre-cancerous condition.

Up-to-date and precise clinical and epidemiological data describing the situation in the Czech Republic is currently unavailable. The Czech Republic still does not have any data on representation of different phenotypes among COPD patients.

The COPD Register is a non-interventional multicenter observational prospective database focusing on the collection and analysis of data on real mortality and morbidity in an unselected (consecutive) population of patients with severe forms of COPD (post-bronchodilator FEV1≤ 60%). Monitoring is done at the occasion of regular check-ups, followed by retrospective search of data in the documentation, and a record into the registry subsequently.

The main purposes of this study:

* Assessment of all-cause mortality
* Assessment of morbidity:

(A) acute exacerbation of COPD (B) acute non-COPD respiratory events (C) acute non-respiratory events (D) cancers (E) ischemic heart disease (infarct, angina pectoris, congestive heart failure and arrhythmia)

Other aims of this study:

* Monitoring of lung function decline (post-bronchodilator FEV1)
* Monitoring of prognostic indices
* COPD categories and quality of life
* Evaluation of activity of daily living
* Assessment of therapeutic compliance

  * Note: MMAS-4 questionnaire by Prof. Donald E. Morisky will not be used as of September 2018
* Analysis of extra-pulmonary impairment during

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilator FEV1/VC < LLN and post-bronchodilator FEV1 ≤ 60% of the predicted value (VC - Vital Capacity, LLN - Lower Limit of Normal)
* Definite clinical diagnosis of COPD (can be overlaps: COPD + asthma / COPD + bronchiectasis)
* Stable course of COPD (≥ 8 weeks free of acute exacerbations and/or free of any acute conditions)
* Informed consent

Exclusion Criteria:

* "Pure" bronchial asthma without COPD
* "Pure" bronchiectasis without COPD
* Cystic fibrosis
* End-stage of COPD
* Non-curable malignancy
* Total non-compliance
* Immobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The COPD registry is a non-interventional multicentre observational prospective database focusing on the collection and analysis of data on real mortality and morbidity in an unselected population of COPD patients in long lasting care of individual participating centres. Each centre covers the population of a certain county. The centres are localized as to symetrically cover the entire Czech Republic.
Sampling Method: Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2013-08; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of all-cause mortality | Outcome measures will be conducted within one year after completion.
  Assessment of all-cause mortality in an unselected group of consecutive patients with severe COPD (post-bronchodilator FEV1 ≤ 60%).

SECONDARY OUTCOMES:
Assessment of morbidity | Outcome measures will be conducted within one year after completion.
  Assessment of morbidity: (A) acute exacerbation of COPD, (B) acute non-COPD respiratory events, (C) acute non-respiratory events, (D) cancers, (E) ischemic heart disease (myocardial infarct, angina pectoris, congestive heart failure and arrhythmia) in an unselected group of consecutive patients with severe COPD (post-bronchodilator FEV1 ≤ 60%).

OTHER OUTCOMES:
Monitoring of lung function decline | Outcome measures will be conducted within one year after completion.
  Monitoring of lung function decline (post-bronchodilator FEV1 will be measured twice a year) and analysis of the differences in patients with specific COPD phenotypes.
Monitoring of activity of daily living | Outcome measures will be conducted within one year after completion.
  Measurement of daily activity using pedometers (each participating patient will be monitored for one month, every year) and analysis of the differences in patients with specific COPD phenotypes.
Monitoring of COPD categories | Outcome measures will be conducted within one year after completion.
  Assessment of the variability in COPD categories (A-D categories will be calculated twice a year) over a 5 year follow-up and analysis of the differences in patients with specific COPD phenotypes.
Monitoring of therapeutic compliance | Outcome measures will be conducted within one year after completion.
  Regular (once a year) monitoring of inhalation technique and evaluation of Morisky Medication Adherence Scale 4 (MMAS-4).
Monitoring of prognostic indices | Outcome measures will be conducted within one year after completion.
  Annual monitoring of several prognostic indices (Celli´s BODE, Puhan´s BODE, ADO) and analysis of the differences in patients with specific COPD phenotypes.
Assessment of the extrapulmonary symptoms | Outcome measures will be conducted within one year after completion.
  Monitoring of the extrapulmonary impairment (Beck depression scale, Zung depression scale, SNOT-22, densitometry, cardiology history, ECG and cardiac ultrasound) and analysis of the differences in subjects with specific COPD phenotypes.
Quality of life assessment(SGRQ) | Outcome measures will be conducted within one year after completion.
  Regular (annual) evaluation of quality of life using SGRQ.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Koblizek, Assoc. Prof. PhD, Principal Investigator — University Hospital Hradec Kralove
Locations (14):
- Czechia (14):
  - University Hospital Brno, Brno
  - Hospital Ceske Budejovice, Ceské Budějovice
  - University Hospital Hradec Kralove, Hradec Králové
  - Hospital Jihlava, Jihlava
  - Regional Hospital Liberec, Liberec
  - Regional hospital Mlada Boleslav, Mladá Boleslav
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - EUC Klinika Plzen, Pilsen
  - Thomayer Hospital, Prague
  - University Hospital in Motol, Prague
  - Hospital Na Bulovce, Prague
  - Masaryk Hospital in Usti nad Labem, Ústí nad Labem
  - Tomas Bata Regional Hospital, Zlín

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Novotna B, Koblizek V, Zatloukal J, Plutinsky M, Hejduk K, Zbozinkova Z, Jarkovsky J, Sobotik O, Dvorak T, Safranek P. Czech multicenter research database of severe COPD. Int J Chron Obstruct Pulmon Dis. 2014 Nov 10;9:1265-74. doi: 10.2147/COPD.S71828. eCollection 2014. PMID 25419124
- [Derived] Brat K, Svoboda M, Hejduk K, Plutinsky M, Zatloukal J, Volakova E, Popelkova P, Novotna B, Engova D, Franssen FME, Vanfleteren LEGW, Spruit MA, Koblizek V. Introducing a new prognostic instrument for long-term mortality prediction in COPD patients: the CADOT index. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2021 Jun;165(2):139-145. doi: 10.5507/bp.2020.035. Epub 2020 Sep 10. PMID 32955038
- See also: Czech National Research Database of COPD — http://chopn.registry.cz/index-en.php